CLINICAL TRIAL: NCT02327338
Title: Use of ThermaCare Heat Wraps and Ibuprofen as an Adjunct to Physical Therapy for Neck Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Future Sciene Technology (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Jerrold Petrofsky, professor, Future Sciene Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A2014
Record Dates: First submitted 2014-12-11; First posted 2014-12-30 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Heat; Pain
MeSH Terms: conditions — Pain | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- continuous low level heat for neck (Experimental): 30 subjects to use ThermaCare heat wraps on their necks for 6 hours before home exercise programs each day for 10 days. Physical therapy 2 times per week will be used on days where heat wraps are not used.
  Interventions: Device: thermacare heat wraps
- Ibuprofen and continuous low level heat (Experimental): 30 subjects to use 1200 mg per day Ibuprofen dosed in 3 dosages 4 hours apart on the same days as heat wraps were to be used. ThermaCare heat wraps to be used on their necks for 6 hours before home exercise programs each day for 10 days. Physical therapy 2 times per week will be used on days where heat wraps and ibuprofen are not used.
  Interventions: Device: thermacare heat wraps; Drug: Ibuprofen
- control (No Intervention): 15 subjects with no heat or ibuprofen just physical therapy 2 times per week.
- sham heat and sham ibuprofen (Sham Comparator): 30 subjects to use 1200 mg per day Ibuprofen sham dosed in 3 dosages 4 hours apart on the same days as sham heat wraps were to be used. ThermaCare heat sham wraps to be used on their necks for 6 hours before home exercise programs each day for 10 days. Physical therapy 2 times per week will be used on days where sham heat wraps andsham ibuprofen are not used.
  Interventions: Device: thermacare heat wraps; Drug: Ibuprofen

INTERVENTIONS:
Device: thermacare heat wraps — off the shelf thermacare continuous heat wraps made by thermacare to produce low level heat on the neck
  Other Names: continuous low level heat
  Arms: Ibuprofen and continuous low level heat; continuous low level heat for neck; sham heat and sham ibuprofen
Drug: Ibuprofen — 1200 mg ibuprofen administered 400mg at 4 hour intervals
  Other Names: advil
  Arms: Ibuprofen and continuous low level heat; sham heat and sham ibuprofen

SUMMARY:
Objective- To see if the use of heat at home between physical therapy sessions results in better therapy outcomes in people with acute neck pain.

Setting: Physical Therapy outpatient rehabilitation center Participants: 90 people with acute nonspecific neck pain broken into 4 groups. Intervention: All subjects will undergo 45 minutes of therapy 2 times per week for 2 weeks. All subjects will accomplish 1 hour of therapeutic exercise at home on days when there is no therapy. Thirty of the subjects will use ThermaCare neck wraps before home exercise, 30 used Ibuprofen plus ThermaCare neck wraps before home exercise, 15 will use a sham heat wrap and an Ibuprofen placebo each day (1200 mg / day) and the last 15 will be controls with conventional physical therapy.

DETAILED DESCRIPTION:
Neck pain patients admitted to an outpatient physical therapy program will be randomly assigned to either a control or 3 experimental groups. An initial evaluation and rehabilitation program will be established which includes a home exercise program. Therapy will be 2 days per week for 2 weeks. Thirty of the subjects will use ThermaCare continuous heat neck wraps applied for 6 hours before home exercise, 30 will use ibuprofen (1200 mg /day given in 3 dosages) plus ThermaCare neck wraps before home exercise, 15 will use a sham heat wrap and a Ibuprofen placebo each day and the last 15 will have conventional therapy. Intervention with heat or Ibuprofen will be used on days that they are not being treated in the clinic. All groups will be evaluated initially and after 2 weeks. They will be given home exercise and heat compliance logs and analog visual pain scales to be filled out each night before exercise and, if they used heat, before and after heat will be applied. The physical therapist will also be asked to evaluate their home compliance, pain and the benefit to them from the heat packs. Subjects will complete a neck disability questionnaire at the beginning and end of the study. At the end of the two weeks of treatment, a multivariate ANOVA will be performed to compare changes in home exercise compliance, functional level, pain level, range of motion, and strength. A statistical level of p≤.05 is considered predictive of a difference between groups.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years

Exclusion Criteria:

* those with neck pain caused by fractures or spinal damage
* those who have undergone neck surgery within the last year
* those with radiculopathy or those with diagnosed diabetes were excluded from this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-11; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
analog visual pain scales | up to 14 days
  subjects will be asked to place a mark on a 10cm line where one end shows no pain and the other represents extreme pain to assess their pain level.

SECONDARY OUTCOMES:
compliance for home exercise | 10 days
  subjects will self assess their compliance for their assigned home exercise program each day of the 10 days they accomplished home exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Iman Khowailed, DSc, Study Chair — Touro University
Locations (1):
- Future Sciecne Technology, Henderson, Nevada, United States